CLINICAL TRIAL: NCT06009744
Title: Effectiveness of Doses of Vitamin c and Zinc in Patients With High Enterocutaneous Fistulas Receiving Nutrition Parenteral Therapy on Closure and Recurrence. Randomized Clinical Trial.
Brief Title: Vitamin C and Zinc in Patients With Enterocutaneous Fistulas.
Acronym: VITAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, ELIZABETH PEREZ CRUZ, MD, MSc, Prof., Hospital Juarez de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HJM 005/32-I
Record Dates: First submitted 2023-07-16; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Enterocutaneous Fistulas
Keywords: enterocutaneous fistulas; Vitamin C; Zinc; Parenteral nutrition
MeSH Terms: conditions — Intestinal Fistula; Hyperphagia | interventions — Ascorbic Acid; Zinc

STUDY DESIGN:
Intervention Model Description: Group a) 25-35 kcal/K/d, 1.3-1.5 g/K/d of amino acids and C 100-300 mg/d y zinc 3-5 mg/d Group b) 25-35 kcal/K/d, 1.3-1.5 g/K/d of amino acids and Vitamin C 1000-2000 mg/d y zinc 10-15 mg/d.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vit C y zinc bajo (Sham Comparator): Parenteral nutrition + Vitamin C 100-300 mg/d y zinc 3-5 mg/d
  Interventions: Drug: Low-dose vitamin C and zinc
- Vit C and zinc alto (Active Comparator): Parenteral nutrition + Vitamin C 1000-2000 mg/d y zinc 10-15 mg/d
  Interventions: Drug: High-dose vitamin C and zinc

INTERVENTIONS:
Drug: Low-dose vitamin C and zinc — This is a randomized, control trial to investigate the effect of Vitamin C and Zinc in patients with enterocutaneous fistulas receiving nutrition parenteral therapy and Vitamin C 100-300 mg/d and zinc 3-5 mg/d
  Other Names: Low Vit C y zinc
  Arms: Vit C y zinc bajo
Drug: High-dose vitamin C and zinc — This is a randomized, control trial to investigate the effect of Vitamin C and Zinc in patients with enterocutaneous fistulas receiving nutrition parenteral therapy and Vitamin C 1000-2000 mg/d y zinc 10-15 mg/d
  Other Names: High Vit C y zinc
  Arms: Vit C and zinc alto

SUMMARY:
Various micronutrients play an important role in the process of closure and recurrence of enterocutaneous fistulas, such as Vitamin C and Zinc. However, there is no specific recommendation on the dose of these nutrients by parenteral route.

DETAILED DESCRIPTION:
This is a randomized, control trial to investigate the effect and safety of doses of vitamin c and zinc in patients with high enterocutaneous fistulas receiving who need nutrition parenteral therapy on closure and recurrence.

Screening will be made to select eligible participants before intervention. Participants were randomly assigned to one of two groups: group a) 25-35 kcal/K/d, 1.3-1.5 g/K/d of amino acids and C 100-300 mg/d y zinc 3-5 mg/d; group b) 25-35 kcal/K/d, 1.3-1.5 g/K/d of amino acids and Vitamin C 1000-2000 mg/d y zinc 10-15 mg/d.

Demographic variables and subjective global assessment scale will be recorded and applied. Anthropometric measurements (weight and body mass index) will be evaluated upon admission and weekly until hospital discharge.

Biochemical markers (albumin, lymphocytes, prealbumin, transferrin, cholesterol, creatinine) and serum metabolic profile (glucose, liver function test) will be measured weekly. During hospitalization, patients will be evaluated daily until the closure of the fistula and/or follow-up at 30 days, monitoring capillary blood glucose, insulin expenditure, and fistula volume.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* >18 years and <70 years old.
* Diagnosis of high-output enterocutaneous fistula for the first time
* Need for parenteral nutrition

Exclusion Criteria:

* Octreotide use
* Palliative care
* Steroid use
* Oxalate nephropathy
* G6PD deficiency
* Hemochromatosis
* Abdominal surgeries in the last 6 months
* Hospitalizations for more than 15 days in the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Fistula closure | follow-up at 30 days
  Evaluate enterocutaneous fistula closure rate.
Recurrence of fistula | follow-up at 30 days
  Evaluate the recurrence of enterocutaneous fistula

SECONDARY OUTCOMES:
Medical-nutritional status | 24-72 hours after hospital admission
  Medical-nutritional status: subjective global assessment
Medical-nutritional status | 24-72 hours after hospital admission
  Medical-nutritional status: nutritional risk index
biochemical markers | every week until a maximum follow-up at 30 days
  Changes in nutritional status biochemical markers: albumin in serum
biochemical markers | every week until a maximum follow-up at 30 days
  Changes in nutritional status biochemical markers: lymphocytes in serum.
biochemical markers | every week until a maximum follow-up at 30 days
  Changes in nutritional status biochemical markers: prealbumin in serum.
biochemical markers | every week until a maximum follow-up at 30 days
  Changes in nutritional status biochemical markers: transferrin in serum.
Metabolic profile | every week until a maximum follow-up at 30 days
  Changes in metabolic profile in serum glucose concentration
Metabolic profile | every 15 days up to a maximum follow-up at 30 days
  Changes in metabolic profile in serum tests liver
Length of hospital stay of patients | follow-up at 30 days
  Determine the length of hospital stay of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Pérez Cruz, Principal Investigator — Hospital Juarez de Mexico
Locations (1):
- Hospital Juárez de México, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeejeebhoy K. Zinc: an essential trace element for parenteral nutrition. Gastroenterology. 2009 Nov;137(5 Suppl):S7-12. doi: 10.1053/j.gastro.2009.08.014. PMID 19874952
- [Background] Yanase F, Fujii T, Naorungroj T, Belletti A, Luethi N, Carr AC, Young PJ, Bellomo R. Harm of IV High-Dose Vitamin C Therapy in Adult Patients: A Scoping Review. Crit Care Med. 2020 Jul;48(7):e620-e628. doi: 10.1097/CCM.0000000000004396. PMID 32404636
- [Background] Couper C, Doriot A, Siddiqui MTR, Steiger E. Nutrition Management of the High-Output Fistulae. Nutr Clin Pract. 2021 Apr;36(2):282-296. doi: 10.1002/ncp.10608. Epub 2020 Dec 24. PMID 33368576
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Background] Girard E, Messager M, Sauvanet A, Benoist S, Piessen G, Mabrut JY, Mariette C. Anastomotic leakage after gastrointestinal surgery: diagnosis and management. J Visc Surg. 2014 Dec;151(6):441-50. doi: 10.1016/j.jviscsurg.2014.10.004. Epub 2014 Oct 22. PMID 25455960